CLINICAL TRIAL: NCT05151185
Title: Establishment of Core Competence and Training Model for Dementia Case Management: Phase 2
Brief Title: Establishment of Core Competence and Training Model for Dementia Case Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Huei-Ling Huang, Associate Professor, PhD, RN, Department of Gerontology and Health Care Management, College of Nursing, Chang Gung University of Science and Technology, Taoyuan, Taiwan, R.O.C, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MOST 110-2511-H-255 -003 -MY2; NMRPF3L0051 (Other: Chang Gung University of Science and Technology)
Record Dates: First submitted 2021-10-31; First posted 2021-12-09 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Dementia
Keywords: dementia; case management; core competence; training program
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The dementia case manager in the control group undergo existing training. The family caregiver in the control group receive routine service.
- training program (Experimental): The dementia case manager in experiment group will undergo training (Competency-based Dementia Case Management Train-the-trainer Program; CDCMTP); The family caregiver in experiment group will receive competency-based Dementia Case Management Service Program.
  Interventions: Other: Case Management Service Program

INTERVENTIONS:
Other: Case Management Service Program — The dementia case manager in experiment group will undergo training (Competency-based Dementia Case Management Train-the-trainer Program; CDCMTP); The family caregiver in experiment group will receive competency-based Dementia Case Management Service Program: Needs Assessment, Intervention, evaluation and follow up, etc. The case management program is provided by a trained case manager in a dementia clinic, as well as telephone consultations and follow-up are provided.
  Arms: training program

SUMMARY:
The purpose of this study is to develop the core competence and training model for case management of dementia. This study is the second phase of the project. The first year is the establishment of the training program and the pilot-test stage. The second year is the project implementation and effectiveness evaluation stage, the intervention effectiveness evaluation of the training course for dementia case managers will be conducted.

DETAILED DESCRIPTION:
The purpose of this study is to develop the core competence and training model for case management of dementia. In the previous year (phase I), the needs and competence assessment stage, the investigators are conducting a survey of the connotation and needs of dementia case management, and explore the role functions and competencies of dementia case managers as the basis for developing the training program.

This study is the second phase of the project. The first year is the establishment of the training program and the pilot-test stage. The data collected in the previous period will be integrated to plan a preliminary training program structure, and then the content and training methods of the training program for dementia case managers will be established using the Delphi method. Then, use this training program to carry out the pilot test of the dementia case managers training program. The second year is the project implementation and effectiveness evaluation stage, the intervention effectiveness evaluation of the training course for dementia case managers will be conducted. The results of this study will serve as a reference for the training program of dementia case managers in future.

ELIGIBILITY:
Inclusion Criteria:

* Dementia Case Managers:

  1. Be at least 20 years old and could communicate in Chinese or Taiwanese.
  2. Currently work for dementia center, dementia care center, or Community-Based Dementia Care Center in Taiwan.
* Dementia family caregivers:

  1. Be at least 20 years old and could communicate in Chinese or Taiwanese.
  2. Primary caregivers
  3. The people with dementia under care are diagnosed with dementia Clinical Dementia Rating Scale(CDR) 0.5 or higher.
  4. Live in northern Taiwan(including Taipei, New Taipei, Taoyuan, and Hsinchu).

Exclusion Criteria:

* Dementia Case Managers:

No longer working for dementia center, dementia care center, or Community-Based Dementia Care Center in Taiwan.

* Dementia family caregivers:

The people with dementia under care live in a long-term care facility or nursing home.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dementia Care Professional Competency Assessment Scale | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline Dementia Care Professional Competency at 1, 3, and 6 months.
  1. The scale was developed by our past research that was supported by the Taiwan Ministry of Science and Technology (Grant Number 106-2511-S-255-002-MY3).
     The scale is used to evaluate dementia care competency in dementia case managers (Huang et al., 2018).
  2. This Scale contains nine subscales (74 items), using Likert 5-point Likert scale from 1 to 5.
     A higher score means better competencies.
  3. This scale is used to evaluate the competence of dementia case managers.
Problem solving, Teamwork Competency Assessment Scale | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline Problem solving, Teamwork Competency at 1, 3, and 6 months.
  1. The scale was developed by our past research that was supported by the Taiwan Ministry of Science and Technology (Grant Number 106-2511-S-255-002-MY3).
     There are 22 questions on this scale. The scale is used to evaluate the problem solving and teamwork competency of Dementia case managers. (Huang et al. 2018).
  2. This scale contains 22 items.10 items were used to evaluate problem solving competencies, 12 items were used to evaluate teamwork competencies.
     A higher score means better competencies.
  3. This scale is used to evaluate the competence of dementia case managers.
Caregiver Preparedness Scale - Professional version | The investigators will evaluate before the intervention, and after intervention for 1, 3, and 6 months. Change from Baseline Caregiver Preparedness - Professional at 1,3, and 6 months.
  1. This scale was developed by our research team by referring to The Preparedness for Caregiving Scale (PCS) developed by Archbold et al.
     This scale is to rate how well prepared they believe they are for caregiving (Archbold et al.,1990; Huang, Kuo, et al., 2013).
  2. This 11-items scale was scored on a 5-point Likert scale from 1 (unprepared) to 5 (well prepared).
     Scores range from 11 to 55, with higher scores representing greater preparedness for caregiving tasks.
     A final question is an open-end question.
  3. This scale is used to evaluate the competence of dementia case managers.
Qualitative interview | The investigators will conduct qualitative interviews after intervention for 1 month. Change from Baseline Qualitative interview at 1 month.
  Conduct qualitative interviews with dementia case managers, focusing on the effectiveness of the training program.
Demographic data of persons with dementia and family caregivers | We will collect demographic data of dementia and family caregivers on the day before the start date of intervention.
  1. The persons with dementia include age, gender, education level, marital status, period of illness, etc.
  2. The family caregivers include age, gender, education level, marital status, etc.
36-item short-form health survey (SF-36) | The investigators will evaluate before the intervention, and after intervention for 1, 3, 6, and 12 months.Change from Baseline 36-item short-form health survey at 1,3,6 and 12 months.
  1. Ware J. E., & Sherbourne, C. D. (1992). The MOS 36-item short-form health survey (SF-36): I.
     Conceptual framework and item selection. Medical care, 473-483.
  2. The SF-36 measures eight scales, with higher scores representing the greater quality of life.
  3. This scale is used to assess the quality of life for people with dementia and their family caregivers .
Dementia Case Management Needs Scale | The investigators will evaluate before the intervention, and after intervention for 1, 3, 6, and 12 months. Change from Baseline Dementia Case Management Needs at 1, 3, 6, and 12 months.
  1. The scale was developed by our past research that was supported by the Taiwan Ministry of Science and Technology (Grant Number 109-2511-H-255-004 -).
     This scale was used to Investigate the needs of case management for family caregivers with dementia in the community.
  2. This Scale uses Likert 5-point Likert scale from 1 to 5, with higher scores representing greater demand for family caregivers.
  3. This scale is used to evaluate family caregivers.
Cohen-Mansfield Agitation Inventory (CMAI) | The investigators will evaluate before the intervention, and after intervention for 1, 3, 6, and 12 months. Change from Baseline behavioral problems (CMAI) at 1, 3, 6, and 12 months.
  1. Dementia's behavioral problems were measured by the Chinese version of the CMAI, community form (Cohen-Mansfield, J et al. 1989, 1991, C.K.Y. Lai, pers. comm.).
  2. The 43-item CMAI has four subscales that assess four groups of behavioral problems: physically non-aggressive behavior, physically aggressive behavior, verbally aggressive behavior and verbally non-aggressive behavior.
     Each item's score ranges from 1 (never happened) to 7 (several times in an hour).
     Scores can range from 43-301, with higher scores representing more frequent or more types of behavioral problems.
  3. This scale is used to evaluate family caregivers.
Agitation Management Self-Efficacy Scale (AMSS) | The investigators will evaluate before the intervention, and after intervention for 1, 3, 6, and 12 months. Change from Baseline caregiver self-efficacy to handle behavioral problems (AMSS) at 1, 3, 6, and 12 months.
  1. Family caregivers' self-efficacy for caring agitated behavior of older people with dementia was measured by the Agitation Management Self-Efficacy Scale (AMSS), which was developed by our research team. (Huang, Shyu, Chen, & Hsu, 2009)
  2. For each of the 43 behavioral problems identified by the Chinese version of the CMAI, caregivers are asked how confident they feel about handling the problem.
     Each AMSS item is scored on a Likert-type scale from 1 (not able to handle at all) to 5 (totally able to handle).
     Total scores range from 43-215. Higher scores represent greater caregiver self-efficacy to handle behavioral problems.
  3. This scale is used to evaluate family caregivers.
Caregiver Preparedness Scale - family caregiver version | The investigators will evaluate before the intervention, and after intervention for 1, 3, 6, and 12 months. Change from Baseline Caregiver Preparedness -family caregiver at 1, 3, 6, and 12 months.
  1. This scale was developed by our research team by referring to The Preparedness for Caregiving Scale (PCS) developed by Archbold et al.
     This scale is to rate how well prepared they believe they are for caregiving (Archbold et al.,1990; Huang, Kuo, et al., 2013).
  2. This 11-items scale was scored on a 5-point Likert scale from 1 (unprepared) to 5 (well prepared).
     Scores range from 11 to 55, with higher scores representing greater preparedness for caregiving tasks.
     A final question is an open-end question.
  3. This scale is used to evaluate family caregivers.
Activities of daily living (ADL) | The investigators will evaluate before the intervention, and after intervention for 1, 3, 6, and 12 months. Change from Baseline ADL at 1, 3, 6, and 12 months.
  1. García-Casal JA, Loizeau A, Csipke E, Franco-Martín M, Perea-Bartolomé MV, Orrell M. Computer-based cognitive interventions for people living with dementia: a systematic literature review and meta-analysis. Aging Ment Health.2016; 25: 1-14.
  2. The ADL refers to activities oriented toward taking care of one's own body.
  3. This scale assesses 10 items related to the activity including feeding, transfer, grooming, toilet use, bathing, mobility, stairs, dressing, bowels, and bladder.
     Each item is scored from 0 (maximum disability and dependency) to 20 (maximum strength and independence).
     Scores can range from 0 to 100, with higher scores representing more independence.
  4. This scale is used to evaluate family caregivers.
Instrumental Activities of Daily Living (IADL) | The investigators will evaluate before the intervention, and after intervention for 1, 3, 6, and 12 months. Change from Baseline IADL at 1, 3 ,6, and 12 months.
  1. Ryu SY, Lee SB, Kim TW, Lee TJ. Subjective memory complaints, depressive symptoms and instrumental activities of daily living in mild cognitive impairment. Int Psychogeriatr. 2015; 11: 1-8.
  2. The IADL refers to activities oriented toward interacting with the environment and that are often complex-generally optional in nature.
  3. This scale assesses 8 items related to the activity including the ability to use a phone, shopping, the model of transportation, meal preparation, housekeeping, laundry, the responsibility for owns medication, and the ability to handle finance.
     Each item is scored from 0 (dependency) to 3 (independence). Scores can range from 0 to 24, with higher scores representing more independence.
  4. This scale is used to evaluate family caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Ling Huang, PhD, Study Chair — Chang Gung University of Science and Technology
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Huang HL, Liao YT, Kung PC, Shyu YL, Hsu WC, Hsu JL. Caregiving management needs and predictors for family caregivers of persons with dementia: a cross-sectional study. BMC Geriatr. 2024 Aug 30;24(1):724. doi: 10.1186/s12877-024-05316-3. PMID 39215257